CLINICAL TRIAL: NCT03332199
Title: A Psycho-educational Intervention for Symptom Cluster Management Among Cancer Patients Undergoing Chemotherapy in Vietnam
Brief Title: A Psycho-educational Intervention for Symptom Cluster Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Ly Nguyen, Principal Investigator, Hanoi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1600000809
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Oncology
Keywords: symptom cluster; oncology; psychoeducation; symptom management; fatigue; pain; sleep disturbance
MeSH Terms: conditions — Neoplasms; Syndrome; Fatigue; Pain; Parasomnias

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group received standard treatment from oncologists and nurses at Hanoi Medical University Hospital.
- Intervention (Experimental): In addition to standard care provided by oncologists and nurses at Hanoi Medical University Hospital as described above, participants assigned to the intervention group received the psychoeducational intervention delivered by the nurse researcher.
  Interventions: Other: Psycho-educational intervention

INTERVENTIONS:
Other: Psycho-educational intervention — The total program, consisting of three intervention sessions, was given over a period of 3 weeks. The one face-to-face session of an-hour's duration was provided within a week of the chemotherapy cycle following recruitment. Two booster sessions of 20-30 minutes were then conducted by phone at one-week intervals after the first intervention session.
  Arms: Intervention

SUMMARY:
The purpose of this study is to develop, implement and undertake a preliminary evaluation of a psychoeducational intervention for managing a cancer-related symptom cluster including pain, fatigue and sleep disturbance experienced by Vietnamese cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Are diagnosed with any type of cancer
* Are over 18 years of age
* Have finished the second chemotherapy cycle
* Expected prognosis of at least 12 months
* Karnofsky level of ≥ 60/100.
* Report three symptoms: fatigue, pain and sleep disturbance at severity level of equal or above 3 during the past 7 days.
* Ability to communicate in Vietnamese

Exclusion Criteria:

* Inability to complete questionnaires or participate in the intervention due to literacy level or communication impairment.
* Have been diagnosed with major psychiatric morbidity such as suicidal tendencies or schizophrenia.

Involved in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Symptom cluster | 4 weeks
  The three-single item Numeric Analogue Scales (fatigue, pain and sleep disturbance) were used at baseline and 4 weeks of the intervention to assess the change of symptom severity at cluster levels. The scales consists of a number of symptoms rated on the 11-point scales, with 0 referring to "not present" and 10 referring to "as bad as you can imagine". The symptom cluster severity was evaluated by averaging symptom summary scores, with a summary higher score indicating greater symptom cluster severity.
Fatigue | 4 weeks
  The Brief Fatigue Inventory (BFI) was used to assess the change of fatigue from baseline to 4 weeks of the intervention. The BFI consists of nine items assessing severity of fatigue in the past 24 hours (4 items) and its impacts on patients' different aspects of life, such as daily activity, emotional well-being, walking ability, work, and social interactions (5 items) on a 11-point scale. A summary higher score indicating greater fatigue severity and interference.
Pain | 4 weeks
  The Brief Pain Inventory was used to assess the change of pain from baseline to 4 weeks of the intervention. The Brief Pain Inventory - Short Form (BPI) encompasses a 4-item pain severity subscale and a 7-item pain interference with daily activities subscale. Each item was rated on 11-point numerical rating scales. A summary higher score indicating greater pain severity and interference.
Sleep disturbance | 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess patients' sleep quality and pattern at baseline and 4 weeks of the intervention. The scale consists of 19 self-reported items categorised in 7 domains, including sleep quality, duration, sleep effectiveness, sleep disturbances, sleep medication, and daytime dysfunction over the last month. Possible scores range from 0 to 21 with a higher score indicating greater sleep disturbance

SECONDARY OUTCOMES:
Performance status | 4 weeks
  Outcome measures included the Karnofsky Performance Scale at baseline and 4 weeks of the intervention. The scale ranges from 10 (moribund, fatal process progressing rapidly) to 100 (normal, no complaints, no evidence of disease).
Depression and Anxiety | 4 weeks
  The Hospital Anxiety and Depression Scale was used to assess the change of depression and anxiety at baseline and 4 weeks of the intervention. The Hospital Anxiety and Depression Scale includes 14 items separated into two subscales for anxiety (HADS-A: 7 items) and depression (HADS-D:7 items). For each sub-scale, the symptom is rated on a 22-point numerical scale which ranges from 0 (no symptom) to 21 (severe).
Health-related quality of life | 4 weeks
  The EQ-5D-5L was used to evaluate health-related quality of life at baseline and 4 weeks of the intervention. The EQ-5D-5L includes five aspects: "mobility, self-care, usual activities, pain/discomfort and anxiety/depression". Each dimension has 5 levels: "no problem, slight problem, moderate problem, severe problem and extreme problem". Possible scores range from 0 to 5 with higher scores indicating poorer quality of five dimensions.
  The EQ VAS records patient's general health-related quality of life on a visual analogue scale, with 0 being "worst imaginable health state" and 100 equal "best imaginable health state".

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen LT, Alexander K, Yates P. Psychoeducational Intervention for Symptom Management of Fatigue, Pain, and Sleep Disturbance Cluster Among Cancer Patients: A Pilot Quasi-Experimental Study. J Pain Symptom Manage. 2018 Jun;55(6):1459-1472. doi: 10.1016/j.jpainsymman.2018.02.019. Epub 2018 Mar 2. PMID 29505795